CLINICAL TRIAL: NCT02782611
Title: Enduring Happiness and Continued Self-Enhancement
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kostadin Kushlev, Postdoctoral Research Associate, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160044
Record Dates: First submitted 2016-04-07; First posted 2016-05-25 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Happiness
Keywords: Happiness; Subjective Well-Being; Psychological Flourishing; Well-Being; Health; Behavioral Change; Life Satisfaction; Affect; Emotion; Goals; Meaning in Life
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): ENHANCE (Enduring Happiness and Continued Self-Enhancement) is a 12-week program that includes an introductory session, 10 weekly sessions focusing on different happiness principles, and a final session focusing on integrating aspects of the program and continuing to practice these principles moving forward. Through completing this program, participants will gain an education on a wide-range of happiness principles and an arsenal of strategies for developing happiness boosting habits and skills.
  Interventions: Behavioral: ENHANCE: Enduring Happiness and Continued Self-Enhancement
- Waiting Group Control (No Intervention): The waiting group control will complete the same assessments as the experimental group but without receiving the intervention.

INTERVENTIONS:
Behavioral: ENHANCE: Enduring Happiness and Continued Self-Enhancement — ENHANCE is a skill-based intervention to teach people a wide variety of strategies that have been shown to boost happiness. Each session of ENHANCE follows a similar format targeted to address three central goals. First, in each session, participants will complete an active learning module designed to educate participants about one of the ten overarching topics featured in this program (e.g., goals, close relationships). Next, participants will engage in activities that put these principles into practice. Finally, this program is designed to encourage a skill-building mindset by helping participants develop habits to integrate these principles into maintained activity in their daily lives moving forward.
  Arms: Treatment

SUMMARY:
Over the past several decades, a new science of subjective well-being has produced insights into the factors that make people happy-from cultivating strong relationships to pursuing the right goals. Drawing on these empirical findings, the investigators created a comprehensive 12-week intervention program, ENHANCE: Enduring Happiness and Continued Self-Enhancement. The investigators multimodal program is designed to teach people essential skills in order to produce sustainable changes in behavior and, as a result, long-lasting increases in happiness. To test the effectiveness of ENHANCE, the investigators designed a six-month randomized clinical trial. Participants will be assigned to an active treatment group or a waiting group control. They will complete baseline assessments, and follow-up assessment at three and six months after the start of the intervention. These assessments will contain measures of subjective well-being and objective measures of health, as well as a variety of psychological mediators (e.g., psychological needs) and moderators (e.g. personality). The investigators will thus be able to explore not only whether ENHANCE works to improve well-being, but also why and how ENHANCE works.

ELIGIBILITY:
Inclusion Criteria:

• Participants ages 25 to 75

Exclusion Criteria:

• Major Depression

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Satisfaction With Life | Baseline, 3, 6 months
  Satisfaction With Life Scale
Change from Baseline in Positive Affect | Baseline, 3, 6 months
  Scale of Positive and Negative Experience: SPANE
Change from Baseline in Negative Affect | Baseline, 3, 6 months
  Scale of Positive and Negative Experience: SPANE
Change from Baseline in Meaning in Life | Baseline, 3, 6 months
  Meaning in Life Questionnaire
Change from Baseline in Thriving | Baseline, 3, 6 months
  Comprehensive Inventory of Thriving

SECONDARY OUTCOMES:
Change from Baseline Positive and Negative Memories Generated by Participants | Baseline, 3, 6 months
  In this task, participants list as many positive (and then negative) life events and then as many negative life events as they can in three minutes. Relative quantities of positive to negative life events that are listed demonstrate accessibility of positive and negative memories, which is an indicator of Subjective Well-Being.
Change from Baseline Peer Reports of Positive Behaviors | Baseline, 3, 6 months
  Peers will be asked to evaluate the participant on how frequently they engaged in a series of affect-related displays over the past week: smiling, laughing,
Change from Baseline Peer Reports of Satisfaction With Life | Baseline, 3, 6 months
Change from Baseline Peer Reports of Positive Affect | Baseline, 3, 6 months
Change from Baseline Peer Reports of Negative Affect | Baseline, 3, 6 months
Change from Baseline Peer Reports of Negative Behaviors | Baseline, 3, 6 months
  Peers will be asked to evaluate the participant on how frequently they engaged in a series of affect-related displays over the past week: crying, frowning, complaining, and criticizing.
Change from Baseline Healthy Behaviors | Baseline, 3, 6 months
  Behavioral Risk Factor Surveillance System
Change from Baseline Perceived Stress | Baseline, 3, 6 months
  Perceived Stress Scale (PSS)
Change from Baseline Depression | Baseline, 3, 6 months
  Patient Health Questionnaire-9
Change from Baseline Self-Esteem | Baseline, 3, 6 months
  Rosenberg Self-Esteem Scale
Change from Baseline Psychological Need Satisfaction: Autonomy, Competence, Relatedness | Baseline, 3, 6 months
  Need Satisfaction Scale
Change from Baseline Body Mass Index: BMI | Baseline, 3, 6 months
Change from Baseline Blood Pressure | Baseline, 3, 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- University of Virginia, Charlottesville, Virginia, United States
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kushlev K, Heintzelman SJ, Lutes LD, Wirtz D, Kanippayoor JM, Leitner D, Diener E. Does Happiness Improve Health? Evidence From a Randomized Controlled Trial. Psychol Sci. 2020 Jul;31(7):807-821. doi: 10.1177/0956797620919673. Epub 2020 Jun 24. PMID 32579432